CLINICAL TRIAL: NCT02425176
Title: A Double-blind Randomised Controlled Trial Investigating the Most Efficacious Dose of Botulinum Toxin-A for Sialorrhoea Treatment in Asian Adults With Neurological Diseases
Brief Title: Botulinum Toxin-A for Sialorrhoea Treatment in Asian Adults With Neurological Diseases
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Mazlina Mazlan, Associate Professor, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UMMC ETHICS 660.1
Record Dates: First submitted 2015-04-09; First posted 2015-04-23 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Sialorrhea
Keywords: botulinum toxin; sialorrhoea; drooling
MeSH Terms: conditions — Sialorrhea | interventions — Botulinum Toxins, Type A; incobotulinumtoxinA; abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Botulinum toxin A (BoNT-A) 50U (Active Comparator): Drug dilution and dosage:
  1. Prepare a mother solution of 500 U/ml by diluting Botulinum toxin A Dysport® with 1 ml of 0.9% saline.
  2. Prepare in 1 ml syringe to get 50U/ml :0.1 ml drawn from the mother solution and add 0.9 ml of 0,9% saline. Total volume of 1 ml.
  Intervention: Botulinum toxin A (BTX-A) 50U are divided equally into 4 salivary glands, 12.5U each gland
  Interventions: Drug: Botulinum toxin A (BoNT-A) 50U
- Botulinum toxin A (BoNT-A) 100U (Active Comparator): Drug dilution and dosage:
  1. Prepare a mother solution of 500 U/ml by diluting Botulinum toxin A Dysport® with 1 ml of 0.9% saline. 2. Prepare in 1 ml syringe to get 100U/ml :0.2 ml drawn from the mother solution and add 0.8 ml of 0.9% saline. Total volume of 1 ml.
  Intervention: Botulinum toxin A (BTX-A) 100U are divided equally into 4 salivary glands, 25U each gland
  Interventions: Drug: Botulinum toxin A (BoNT-A) 100U
- Botulinum toxina A (BoNT-A) 200U (Active Comparator): Drug dilution and dosage:
  1. Prepare a mother solution of 500 U/ml by diluting Botulinum ToxinA Dysport® with 1 ml of 0.9% saline. 2. Prepare in 1 ml syringe to get 200U/ml :0.4 ml is drawn from the mother solution and 0.6ml of 0.9% saline is added. Total volume of 1 ml.
  Intervention: Botulinum toxin A (BTX-A) 200U are divided equally into 4 salivary glands, 50U each gland
  Interventions: Drug: Botulinum toxin A (BoNT-A) 200U

INTERVENTIONS:
Drug: Botulinum toxin A (BoNT-A) 50U — Drug intervention:
  The total dose is divided equally and injected into 4 salivary glands (submandibular and parotid gland bilaterally) via a 25G or 23G needle with ultrasound guidance. One site is injected per gland.
  Drug is only injected once at baseline
  Other Names: Dysport
  Arms: Botulinum toxin A (BoNT-A) 50U
Drug: Botulinum toxin A (BoNT-A) 100U — The total dose is divided equally and injected into 4 salivary glands (submandibular and parotid gland bilaterally) via a 25G or 23G needle with ultrasound guidance. One site is injected per gland.
  Other Names: Dysport
  Arms: Botulinum toxin A (BoNT-A) 100U
Drug: Botulinum toxin A (BoNT-A) 200U — The total dose is divided equally and injected into 4 salivary glands (submandibular and parotid gland bilaterally) via a 25G or 23G needle with ultrasound guidance. One site is injected per gland.
  Other Names: Dysport
  Arms: Botulinum toxina A (BoNT-A) 200U

SUMMARY:
The efficacy of Botulinum toxin A (BoNT-A) in Asian population has not been properly studied and there is no literature available on the most efficacious dose of BoNT-A for sialorrhoea treatment. This research is aimed to find the dose of Dysport® that would be efficacious without treatment-related adverse events and the duration of effectiveness of the drug for sialorrhea treatment in Malaysian patients. The efficacy, safety, tolerability and adverse effects of three doses of Dysport®(50MU, 100MU and 200MU) are examined at 2,6,12 and 24 weeks post injection in this double-blinding, randomized trial.

DETAILED DESCRIPTION:
Study Objectives:

To determine the efficacy, safety, tolerability and adverse effects of three doses of Dysport® (50MU, 100MU and 200MU) in the treatment of sialorrhoea in Asian patients with neurological disorders/diseases and to determine the most efficacious dose.

Study design:

Dose-ranging double blind pilot study.

Sample size:

At least 30 adult patients with various neurological disorders complicated with sialorrhoea including stroke, motor neurone disease, traumatic brain injury and Parkinsonism would be divided into 3 dosing groups.

Study method:

Patients who satisfy inclusion criteria and have given informed consent would be randomized into 3 equal groups given different total doses-50MU, 100MU, 200MU. The total dose will be divided equally and give to each of 4 salivary glands viz. the submandibular and parotid gland bilaterally. For example, if 200MU is to be given in total, 50MU would be given to each gland. Injections would be given via a 25G needle to each gland with ultrasound guidance for better needle placement. One site will be injected per gland.

Primary outcome measure The percentage reduction in the rate of saliva production (as measured by difference in mean weight of dental rolls per minute from baseline) for each of the groups given different doses of Dysport® at 2,6,12 and 24 weeks post injection.

Secondary outcome measure

1. Patient's subjective assessment of improvement in sialorrhoea using the Drooling Frequency and Severity Scale (Thomas-Stonell scale) at 2,6,12 and 24 weeks post-injection.
2. Duration to maximum reduction in salivation (as measured by the maximum reduction in weight of dental rolls)

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years old.
2. Patients with neurological disorder including stroke, motor neurone disease, traumatic brain injury and Parkinsonism, diagnosis confirmed clinically by their treating physicians.
3. Patients with a Thomas-Stonell Drooling Frequency and Severity Scale combined drooling ranking of ≥5.
4. Patients who are able to give signed informed consent and are willing and able to comply with scheduled visits, treatment plan and other study procedure.

Exclusion Criteria:

1. Patients who are pregnant.
2. Patients with bleeding disorders or who are on anticoagulants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-09; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the amount of saliva produced within 6 months | 2,6,12 and 24 weeks post injection
  the amount of saliva produced was measured by the differential weight of a dental roll gauze placed in the buccal mucosal cavity calculated via an electronic microbalance scale to the nearest 0.0001 g

SECONDARY OUTCOMES:
subjective report of sialorrhea/ drooling within 6 months post injection | 2,6,12 and 24 weeks post injection
  subjective report of sialorrhea using the Drooling Frequency and Severity Scale (DFS).

CONTACTS AND LOCATIONS:
Overall Officials: MAZLINA MAZLAN, MBBS, MRM, Principal Investigator — University of Malaya; SAINI ABDULLAH, MBBS, MRM, Study Chair — KPJ KL REHABILITATION CENTRE
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, W.persekutuan, Malaysia